CLINICAL TRIAL: NCT05207774
Title: Pre-operative Intranasal Oxytocin for Enhancing Bariatric-induced Diabetes remissionPre-operative Intranasal Oxytocin for Enhancing Bariatric-induced Diabetes Remission
Brief Title: Pre-operative Intranasal Oxytocin for Enhancing Bariatric-induced Diabetes Remission
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOR-0041-18-CTIL
Record Dates: First submitted 2019-10-23; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Obesity; Diabetes; Bariatric Surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin (Experimental): 8 U/oxytocin three-times daily, 30 min before breakfast, lunch and dinner, using a nasal atomizer for 8 weeks
  Interventions: Drug: Oxytocin
- placebo (Placebo Comparator): intranasal spray containing placebo three-times daily, 30 min before breakfast, lunch and dinner, using a nasal atomizer for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Oxytocin — 8 weeks intranasal oxytocin 24 units per day. 8 units prior each meal. 4units/0.1 ml per puff
  Arms: oxytocin
Drug: placebo — 8 weeks intranasal placebo 0.6 ml per day. . 0.1 ml per puff
  Arms: placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled study of the effects of intranasal oxytocin in obese adults with diabetes undergoing bariatric surgery. Subjects will be randomized to receive of intranasal oxytocin or placebo (8 units 3 times daily) for 8 weeks prior surgery. Study visits include screening to determine eligibility, CGM will be connected before and after oxytocin administration, and 1 year post surgery. blood tests including oral glucose tolerance test will be done and fat samples will be taken during surgery. The investigator's hypothesis is that oxytocin administration prior bariatric surgery can induce diabetes remission in patients with diabetes

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Diabetes Mellitus type 2
* HBA1C < or= 9
* BMI >35
* eligible for bariatric surgery (after a hospital bariatric committee)
* Advanced diarem>6
* Signed an informed consent -

Exclusion Criteria:

* HBA1C above 9
* Prior bariatric surgery in the past 6 years
* secondary diabetes
* steroid therapy
* uncontrolled hypertension(>180/100)
* Arythmia: paroxysmal tachyarythmia or high degree AV-Block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with diabetes remission 1 year post surgery | 1 year post surgery
  HBA1C less then 6.5% without need for diabetes medication
Number of participants who improved their glycemic control | 8 weeks
  increase in "Time in Range" by 10% and or decrease in HBA1C by 1 % 8 weeks from treatment
weight loss | 8 weeks
  weight reduction - kg.
weight loss | 1 year
  weight reduction - kg.
obesity | 8 weeks
  change in waist circumference
obesity | 1 year
  change in waist circumference

SECONDARY OUTCOMES:
Rate of Insulin secretion | 8 weeks
  Increase of insulin secretion after oxytocin administration
Rate of Insulin secretion | 1 year
  Increase of insulin secretion after oxytocin administration
Rate of insulin resistance | 8 weeks
  Increase of insulin sensitivity after oxytocin administration
Rate of insulin resistance | 1 year
  Increase of insulin sensitivity after oxytocin administration
lipids-LDL CHOLESTEROL | 8 weeks
  change in lipid profile: LDL
lipids-LDL CHOLESTEROL | 1 year
  change in lipid profile: LDL
lipids-HDL CHOLESTEROL | 8 weeks
  change in lipid profile: HDL
lipids-HDL CHOLESTEROL | 1 year
  change in lipid profile: HDL
lipids-NON HDL CHOLESTEROL | 8 weeks
  change in lipid profile: NON HDL cholesterol. triglycerides
lipids-NON HDL CHOLESTEROL | 1 year
  change in lipid profile: NON HDL cholesterol. triglycerides
lipids-Triglycerides | 8 weeks
  change in lipid profile: triglycerides
lipids-Triglycerides | 1 year
  change in lipid profile: triglycerides
blood pressure | 8 weeks
  change in systolic and diastolic blood pressure
blood pressure | 1 year
  change in systolic and diastolic blood pressure
urine microalbumin | 8 weeks
  Change in microalbumin/creatinin
urine microalbumin | 1 year
  Change in microalbumin/creatinin
HPA axis | 8 weeks
  change in cortisol
HPA axis | 1 year
  change in cortisol
HPA axis | 8 weeks
  change in ACTH
HPA axis | 1 year
  change in ACTH
systemic inflammation | 8 weeks
  changes of inflammation markers: hrCRP
systemic inflammation | 1 year
  changes of inflammation markers: hrCRP
systemic inflammation | 8 weeks
  changes of inflammation markers: IL-6
systemic inflammation | 1 year
  changes of inflammation markers: IL-6
systemic inflammation | 8 weeks
  changes of inflammation markers: TNFα
systemic inflammation | 1 year
  changes of inflammation markers: TNFα
systemic inflammation | 8 weeks
  changes of inflammation markers: IL-1α
systemic inflammation | 1 year
  changes of inflammation markers: IL-1α
systemic inflammation | 8 weeks
  changes of inflammation markers: IL-1RA
systemic inflammation | 1 year
  changes of inflammation markers: IL-1RA
systemic inflammation | 8 weeks
  changes of inflammation markers: IL-17
systemic inflammation | 1 year
  changes of inflammation markers: IL-17
systemic inflammation | 8 weeks
  changes of inflammation markers: IL-21
systemic inflammation | 1 year
  changes of inflammation markers: IL-21
systemic inflammation | 8 weeks
  changes of inflammation markers: adiponectin
systemic inflammation | 1 year
  changes of inflammation markers: adiponectin
systemic inflammation | 8 weeks
  changes of inflammation markers: leptin
systemic inflammation | 1 year
  changes of inflammation markers:leptin
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: E2F1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: ASK1/2
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: LC3-II
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: family of ATGs
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated:p-62
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: TRAL
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: TL-1A
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: CCL5
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated:RB1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated:LEPTIN.
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: CCL2,
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated:CCL8
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated:CD68
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: BECN1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: TFDP1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: ADIPOQ,
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: NCK2
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: TP53
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: COL6A1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: COL3A1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: KIT
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: CMA1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: RIPK1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated:TNF
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: CD36
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: IL-6
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: ELN
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: CD11C
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated:CD206
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: CD163
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: CD209
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: CTGF
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: PEPD
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: PAI-1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: BCKDHB
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated:HADHA
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: MMUT
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: ALDH6A1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: endogenous control-PGK1
omental and subcutaneous fat inflammation | 8 weeks
  Real time PCR - mRNA will be extracted, cDNA will be generated and the following genes will be evaluated: endogenous control PPIA
omental and subcutaneous fat inflammation | 8 weeks
  Western blot analysis -The following proteins will be evaluated: E2F1
omental and subcutaneous fat inflammation | 8 weeks
  Western blot analysis -The following proteins will be evaluated: ASK1
omental and subcutaneous fat inflammation | 8 weeks
  Western blot analysis -The following proteins will be evaluated: p-62
omental and subcutaneous fat inflammation | 8 weeks
  Western blot analysis -The following proteins will be evaluated: TRAL
omental and subcutaneous fat inflammation | 8 weeks
  Western blot analysis -The following proteins will be evaluated: TL-1A,
omental and subcutaneous fat inflammation | 8 weeks
  Western blot analysis -The following proteins will be evaluated: PEPD
omental and subcutaneous fat inflammation | 8 weeks
  Western blot analysis -The following proteins will be evaluated: PAI-1
omental and subcutaneous fat inflammation | 8 weeks
  Western blot analysis -The following proteins will be evaluated: family of ATGs
omental and subcutaneous fat inflammation | 8 weeks
  Western blot analysis -The following proteins will be evaluated: endogenous control -beta-actin
omental and subcutaneous fat inflammation | 8 weeks
  ELISA: adiponectin
omental and subcutaneous fat inflammation | 8 weeks
  ELISA: leptin
omental and subcutaneous fat inflammation | 8 weeks
  ELISA: TNF
omental and subcutaneous fat inflammation | 8 weeks
  ELISA: IL-6
omental and subcutaneous fat inflammation | 8 weeks
  histological studies :Adipocyte size distribution.
omental and subcutaneous fat inflammation | 8 weeks
  histological studies : CD68 staining
omental and subcutaneous fat inflammation | 8 weeks
  histological studies :,c-kit staining
omental and subcutaneous fat inflammation | 8 weeks
  Culture of explants in media for up to 1 week for obtaining medium with secreted products of the tissue. Following secreted products will be measured using ELISA: adiponectin
omental and subcutaneous fat inflammation | 8 weeks
  Culture of explants in media for up to 1 week for obtaining medium with secreted products of the tissue. Following secreted products will be measured using ELISA: leptin
omental and subcutaneous fat inflammation | 8 weeks
  Culture of explants in media for up to 1 week for obtaining medium with secreted products of the tissue. Following secreted products will be measured using ELISA: TNF
omental and subcutaneous fat inflammation | 8 weeks
  Culture of explants in media for up to 1 week for obtaining medium with secreted products of the tissue. Following secreted products will be measured using ELISA: IL-6
omental and subcutaneous fat inflammation | 8 weeks
  Culture of explants in media for up to 1 week for obtaining medium with secreted products of the tissue. Following secreted products will be measured using ELISA: CTRP6/12/2 (ng/ml).

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka Unuversity Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Yes